CLINICAL TRIAL: NCT07099612
Title: Usability and Feasibility of a Smart Blister System With and Without a Mobile App: A Mixed-Methods Study
Brief Title: Smart Blister Packaging and Mobile Application to Monitor and Support Medication Adherence: a Two-arm Usability Study
Acronym: SMART-BLISTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Aardex Group (Unknown); Smurfit Westrock (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18348
Record Dates: First submitted 2025-05-20; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer Study
Keywords: smart blister; medication intake; medication monitoring; adherence; digital health; medication compliance; self-management; patient behavior; usability; feasibility; user experience; System Usability Scale; mixed-methods; pilot
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment design with two arms. Participants are randomly assigned to one of two groups in a 1:1 ratio at the start of the study and remain in their assigned group for the entire 8-week study period.
  Arm 1 (Intervention Group): Participants use the Cere®Pak smart blister system in combination with the MEMS® Mobile smartphone application. The app provides optional reminders, access to dosing history, and allows users to manually edit or confirm recorded dose events.
  Arm 2 (Control Group): Participants use the Cere®Pak smart blister system without the MEMS® Mobile app. This group receives no digital reminders or adherence feedback during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Blister System + MEMS® Mobile App (Experimental): Participants in this group will use the Cere®Pak smart blister system in combination with the MEMS® Mobile smartphone application. The app connects to the blister pack via near-field communication (NFC) and provides optional reminder notifications, visual feedback on adherence history, and the ability to manually edit or confirm dose events. Participants will use the system for 8 weeks, following a simulated twice-daily medication schedule using placebo tablets. Tablets are not ingested. Adherence data is recorded electronically and synchronized through the app.
  Interventions: Device: MEMS® Mobile smartphone application; Device: Cere®Pak smart blister pack
- Smart Blister System Only (No App) (Active Comparator): Participants in this group will use the Cere®Pak smart blister system without access to the MEMS® Mobile app or its features. The smart blister electronically records tablet removal, but participants do not receive reminders or adherence feedback. They will follow the same 8-week, twice-daily placebo schedule as the intervention group. Tablets are not ingested. This group serves as a control to assess the added value of the app in terms of usability and adherence.
  Interventions: Device: Cere®Pak smart blister pack

INTERVENTIONS:
Device: MEMS® Mobile smartphone application — The MEMS® Mobile app is a smartphone application that connects to the Cere®Pak smart blister pack via near-field communication (NFC). It allows participants to view their medication intake history, receive optional reminders, and manually edit or confirm recorded dosing events. The app is installed on the participant's own smartphone (iOS or Android) and used throughout the 8-week study period. Participants are encouraged to scan their blister at least once daily to synchronize data. This intervention is for the Arm 1 group only.
  Arms: Smart Blister System + MEMS® Mobile App
Device: Cere®Pak smart blister pack — The Cere®Pak is an electronic blister pack with 28 cavities containing placebo tablets. It automatically records the date and time when each cavity is opened, using embedded electronics. Participants are instructed to simulate a twice-daily medication schedule (morning and evening) for 8 weeks by pushing out tablets without ingesting them. The device functions independently in the control group and connects with the MEMS® Mobile app in the intervention group. Both arms work with this intervention.

SUMMARY:
Many people struggle to take their medications as prescribed, which can lead to poor health outcomes and increased healthcare costs. New technologies, such as smart blister packs and mobile apps, may help patients improve how they take their medicine. These systems can record when a tablet is taken and give reminders or feedback through a smartphone.

This study evaluates the usability and feasibility of a smart medication packaging system called Cere®Pak, which automatically logs each time a tablet is removed. A connected mobile application, MEMS® Mobile, can provide additional support such as reminders and dose tracking.

The goal of this study is to compare the user experience of the Cere®Pak system with and without the use of the app. We hypothesize that participants using the app in addition to the smart blister will report better usability and may show higher engagement with the system.

The study is a small, randomized trial involving healthy adult volunteers. Participants are randomly assigned to one of two groups: One group uses the Cere®Pak system together with the MEMS® Mobile app, which includes optional reminders and access to adherence data. The other group uses the Cere®Pak system alone, without the app or digital feedback.

Participants are asked to simulate taking a placebo tablet twice daily for eight weeks by pushing tablets out of the blister pack (without ingesting them). The study measures usability through questionnaires, medication-taking behavior through electronic monitoring and pill counts, and collects feedback through short interviews.

This study will help determine how acceptable and usable this technology is, and whether the mobile app adds value in supporting consistent medication use.

DETAILED DESCRIPTION:
This randomized controlled pilot study investigates the usability and feasibility of the Cere®Pak smart blister system, with and without integration of the MEMS® Mobile smartphone application, in healthy adult volunteers. The study evaluates whether the addition of a mobile app improves the user experience and adherence behavior compared to the use of the smart blister pack alone.

Cere®Pak is an electronic blister system that automatically logs the date and time of each dose dispensed. The MEMS® Mobile app connects with the blister pack via near-field communication (NFC), enabling users to receive reminders, view their adherence data, and manually edit dosing events if needed. The app is compatible with iOS and Android smartphones and allows users to activate or deactivate features such as notifications and data visualization.

Participants are randomized in a 1:1 ratio into two parallel arms:

* Intervention Group (Arm 1): participants use the Cere®Pak system in combination with the MEMS® Mobile app.
* Control Group (Arm 2): participants use the Cere®Pak system without app support (i.e., no reminders or adherence feedback).

The study runs over an 8-week period. Participants receive four 28-count placebo blister packs, simulating a twice-daily medication regimen. They are instructed to push out tablets at the designated times, but not to ingest them. Data on blister openings are recorded electronically. App users are instructed to scan the pack regularly to synchronize data.

Primary outcomes include: The System usability, assessed via the System Usability Scale (SUS), a 10-item validated questionnaire. Additionally, qualitative user feedback collected via semi-structured interviews.

Secondary outcomes include: Medication adherence based on electronic records (raw and adjusted for technical malfunctions). Secondly, adherence verification via manual pill counts at the end of the follow-up period. Finally, app usage data (e.g., scan frequency, use of editing function, reminder engagement).

The study also includes technical performance monitoring. Device malfunctions (e.g., battery failures, sensor disconnection) are logged and excluded from adherence calculations when relevant.

This trial uses a mixed-methods approach to evaluate both objective outcomes and subjective user experience. The results will inform future implementation of smart medication packaging systems and the role of app-based feedback in promoting adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to read and understand English
* Owns a compatible smartphone (iOS version ≥13 or Android version ≥8)
* Willing and able to use a smart blister pack system for 8 weeks
* Provides informed consent

Exclusion Criteria:

* Severe physical or cognitive limitations that interfere with the use of blister packaging or smartphone apps
* Known allergy or sensitivity to the materials in the blister packaging (even though tablets are not ingested)
* Serious health conditions that significantly limit daily functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
System Usability Score (SUS) | Week 8 (end of study participation)
  Usability of the smart blister system will be assessed using the System Usability Scale (SUS), a validated 10-item questionnaire measuring perceived ease of use, effectiveness, and satisfaction. Participants in both study arms will complete the SUS at the end of the 8-week study period. Units: Score from 0 to 100 (higher = better usability)
Qualitative User Experience Feedback | Week 8
  Participants will complete a semi-structured interview at the end of the study to explore their experience using the smart blister system, perceived usefulness, ease of integration into daily life, and suggestions for improvement. Transcripts will be analyzed thematically.

SECONDARY OUTCOMES:
Medication Adherence (Digital Measurement) | Cumulative over the 8-week study period
  Medication adherence will be calculated as the proportion of scheduled doses registered by the smart blister system. Days with device malfunction will be excluded from analysis. Adherence will be expressed as the percentage of recorded doses versus expected doses over 8 weeks. Units: Percentage (%).
Medication Adherence (Manual Pill Count) | Week 8 (final visit)
  Adherence will also be assessed through manual pill counts of returned blister packs at the final study visit. The number of tablets removed will be compared to the expected number over the 8-week study period. Units: Number of tablets taken / Percentage (% adherence)
App Usage - Number of Blister Scans | Cumulative over 8 weeks
  Total number of times the participant scanned the blister pack using the MEMS® Mobile app. Unit: Count (n)
App Usage - Number of Manually Edited Doses | Cumulative over 8 weeks
  Total number of doses that were manually edited or confirmed by the participant. Unit: Count (n)
App Usage - Days with App Interaction | Cumulative over 8 weeks
  Description: Number of days during the 8-week study period on which the participant interacted with the app. Unit: Number of Days

OTHER OUTCOMES:
Exploratory Subgroup Analyses of Usability (SUS) scores | Week 8
  Comparison of mean SUS scores across predefined subgroups, including age, gender, and prior experience with medication use. Unit: SUS Score (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Job F.M. van Boven, PharmD, PhD, Principal Investigator — Department of Clinical Pharmacy & Pharmacology, University Medical Center Groningen (UMCG), University of Groningen, Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD) due to the small sample size, the non-clinical nature of the data, and privacy considerations. The study was conducted as a pilot usability evaluation, and the primary outcomes do not involve sensitive health data or clinical endpoints. While individual-level data may be made available upon reasonable request in the future, there is no formal data sharing plan in place at this time.